CLINICAL TRIAL: NCT06718374
Title: Chest Pain Symptoms Differences Between Diabetes Mellitus and Non-diabetes Mellitus Patients with Acute Coronary Syndrome
Brief Title: Chest Pain Symptoms Differences Between Diabetic Patients and Non
Acronym: chestpaindm
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Antonios Samir Ishak Ibrahim, assiut hospital, Assiut University
Other Study IDs: chestpain
Record Dates: First submitted 2024-07-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chest Pain; Diabetes Mellitus
MeSH Terms: conditions — Chest Pain; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- non diabetic
- diabetic

SUMMARY:
Cardiovascular disease is the most severe cause of death among all non-infectious diseases and accountable for 17.5 million deaths in the world. Heart mortality in patients with DM is frequently associated with prevalence silent ischemia, which is triggered by autonomic neuropathy, thereby decreasing the chest pain felt by them

ELIGIBILITY:
Inclusion Criteria:

i) Patients diagnosed with STEMI and NSTEMI ii) Both genders iii) above the age of 30 years iv) Patients with acute myocardial infarction with or without chest pain (angina) for 24 hours v) patients who are hemodynamically stable vi) patients without acute decompensated heart failure (ADHF) vii) patients without malignant arrhythmias viii) patients without in Acute Lung Oedem (ALO) condition ix) patients not using ventilator x) patient willing to and become respondents.

Exclusion Criteria:

i) Patients with several complications, thereby making it impossible to interview them ii) patients who have never undergone CABG surgery iii) patients who refuse to be respondents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases admitted to ED who meet the eligibility criteria will be recruited in this study after obtaining an informed consent chest pain of DM and non-DM patients with the acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hospital admission | 1 day
Intensive Care Unit admission | One week
Mortality | One month

CONTACTS AND LOCATIONS:
Overall Officials: Essam El-dien M Abdullah, MD, Study Director — Assiut University; Zeinab Abd-Elatiff, MD, Study Director — Ismailia Universiry; Khalid Abdelbaky, MD, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No